CLINICAL TRIAL: NCT05800145
Title: Pilot Study to Evaluate the Feasibility of Using a Sequential Multiple Assignment Randomized Trial to Address Food Insecurity in Patients With Hypertension (Pilot SMART-FI)
Brief Title: Trial to Address Food Insecurity in Patients With Hypertension (SMART-FI)
Acronym: SMART-FI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00094934; 5K23HL146902-04 (NIH)
Record Dates: First submitted 2023-03-22; First posted 2023-04-05 (Actual); Results first posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2024-09

CONDITIONS: Hypertension
Keywords: Food Insecurities; Systolic Blood Pressure; cardiovascular disease
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — Community Health Workers

STUDY DESIGN:
Intervention Model Description: The objective of this study is to conduct a pilot sequential multiple assignment randomized trial (SMART) addressing food insecurity in patients with uncontrolled Hypertension (HTN) to determine the feasibility of recruitment/retention and the potential impact on blood pressure in anticipation of a larger more definitive trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- resource referral (Experimental): will receive a tailored list of information about community resources. The list will include information about local emergency food resources (e.g. local food pantries) and government programs to address Food Insecurities (FI) Supplemental Nutrition Assistance Program (SNAP).
  Interventions: Behavioral: Resource information Supplemental Nutrition Assistance Program (SNAP)
- community health worker (CHW) intervention (Active Comparator): assist participants in addressing FI and supporting them in their blood pressure management
  Interventions: Behavioral: community health worker (CHW)
- medically tailored meals (MTM) (Active Comparator): Participants will receive 10 medically tailored meals delivery to their home weekly for 3 months
  Interventions: Behavioral: medically tailored meals

INTERVENTIONS:
Behavioral: Resource information Supplemental Nutrition Assistance Program (SNAP) — Participants randomized to the resource referral arm will receive a tailored list of information about community resources. The list will include information about local emergency food resources (e.g. local food pantries) and government programs to address FI (e.g. SNAP).
  Other Names: SNAP
  Arms: resource referral
Behavioral: community health worker (CHW) — Participants randomized to the CHW intervention will have an initial baseline visit scheduled at a mutually convenient location.
  Other Names: CHW
  Arms: community health worker (CHW) intervention
Behavioral: medically tailored meals — Participants will receive 10 medically tailored meals delivery to their home weekly for 3 months
  Other Names: MTM
  Arms: medically tailored meals (MTM)

SUMMARY:
In the US, 47% of adults have hypertension (HTN), and HTN accounts for more cardiovascular disease (CVD) deaths than any other CVD risk factor. Thus, the lack of an adaptive, stepped-care intervention to address FI in patients with HTN is a critical problem affecting a large, vulnerable population.

DETAILED DESCRIPTION:
Despite advances in prevention and treatment, barriers to adherence are common and HTN disparities remain pervasive. Populations that have been socially and economically disadvantaged have a greater prevalence of HTN, worse blood pressure control, and are at higher risk of developing CVD from HTN. Food insecurity (FI), the lack of consistent access to nutritionally adequate foods, is an important social need that affects 30 million people in the US, impacts adherence to treatment, and contributes to HTN disparities. Increasingly, health systems are investing in interventions to address FI as part of routine care, including lower-cost, low intensity (e.g. providing information about community resources) and higher-cost, high intensity (e.g. using community health workers (CHWs), delivery of medical tailored meals (MTM)) interventions

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years of age)
* diagnosis of Hypertension (HTN) (defined by ICD-10 code) or have been prescribed at least one blood pressure medication (including thiazide diuretic, calcium channel blocker, beta-blocker, angiotensin-converting enzyme inhibitors, or angiotensin receptor blocker)
* blood pressures at their primary care office was >130/80
* experience Food Insecurity (FI) based on the 2-item Hunger Vital Sign
* live in Winston-Salem or Forsyth County

Exclusion Criteria:

* unable to speak English or Spanish
* have severe cognitive impairment or major psychiatric illness that prevents consent and participation
* lack of safe, stable residence and ability to store meals
* pregnant, breastfeeding, or planning to become pregnant in the next year
* advance kidney disease (estimated creatine clearance < 30 mL/min)
* serious medical condition which either limits life expectancy or requires active management
* those planning on moving out of the geographic area within 12 months
* lack of a telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Palakshappa, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant data that underlie the Results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose

RESULTS

PARTICIPANT FLOW:
Groups:
- Resource Referral Only: This arm included participants who responded to resource information in Stage 1 and participants who were not assessed for response at the end of Stage 1. In Stage 1, participants received a tailored list of information about community resources. The list will include information about local emergency food resources (e.g. local food pantries) and government programs to address Food Insecurity (FI), such as the Supplemental Nutrition Assistance Program (SNAP).
  In Stage 2, responders did not receive any additional intervention than the information provided in Stage 1.
- Resource Referral + CHW: This arm includes participants who did not respond to resource information in Stage 1. In Stage 1, participants received a tailored list of information about community resources. The list will include information about local emergency food resources (e.g. local food pantries) and government programs to address Food Insecurity (FI), such as the Supplemental Nutrition Assistance Program (SNAP).
  In Stage 2, nonresponders to resource information received assistance from a community health worker (CHW) for 3 months. The CHW helped participants with accessing community resources and worked directly with the patient's care team to assist with any barriers to care.
- Resource Referral + Medically Tailored Meals (MTM): This arm included participants who did not respond to resource information in Stage 1. In Stage 1, participants received a tailored list of information about community resources. The list will include information about local emergency food resources (e.g. local food pantries) and government programs to address Food Insecurity (FI), such as the Supplemental Nutrition Assistance Program (SNAP).
  In Stage 2, nonresponders received 10 medically tailored meals delivered to their home weekly for 3 months.
- Community Health Worker (CHW) Only: This arm included participants who responded to resource information in Stage 1 and participants who were not assessed for response at the end of Stage 1. In Stage 1, participants received assistance from a community health worker (CHW) for 3 months. The CHW helped participants with accessing community resources and worked directly with the patient's care team to assist with any barriers to care.
  In Stage 2, responders did not receive any additional intervention than the CHW assistance provided in Stage 1.
- Community Health Worker (CHW) + CHW Assitance: This arm includes participants who did not respond to CHW assistance in Stage 1. In Stage 1, participants received assistance from a CHW for 3 months. The CHW helped participants with access community resources and worked directly with the patients care team to assist with any barriers to care.
  In Stage 2, nonresponders to CHW assistance in Stage 1 received assistance from a CHW for an additional 3 months.
- Community Health Worker (CHW) Assistance + Medically Tailored Meals (MTM): This arm includes participants who did not respond to CHW assistance in Stage 1. In Stage 1, participants received assistance from a CHW for 3 months. The CHW helped participants with access community resources and worked directly with the patients care team to assist with any barriers to care.
  In Stage 2, nonresponders received 10 medically tailored meals delivered to their home weekly for 3 months.
Period: Stage 1 Intervention (Months 1-3)
Arm/Group | Resource Referral Only | Resource Referral + CHW | Resource Referral + Medically Tailored Meals (MTM) | Community Health Worker (CHW) Only | Community Health Worker (CHW) + CHW Assitance | Community Health Worker (CHW) Assistance + Medically Tailored Meals (MTM)
Started | 13 | 7 | 8 | 18 | 6 | 8
Completed | 5 | 7 | 8 | 12 | 6 | 8
Not Completed | 8 | 0 | 0 | 6 | 0 | 0
Not completed — Lost to Follow-up | 7 | 0 | 0 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 3 | 0 | 0
Period: Stage 2 Intervention (Months 4-6)
Arm/Group | Resource Referral Only | Resource Referral + CHW | Resource Referral + Medically Tailored Meals (MTM) | Community Health Worker (CHW) Only | Community Health Worker (CHW) + CHW Assitance | Community Health Worker (CHW) Assistance + Medically Tailored Meals (MTM)
Started | 5 | 7 | 8 | 12 | 6 | 8
Completed | 4 | 2 | 8 | 9 | 4 | 7
Not Completed | 1 | 5 | 0 | 3 | 2 | 1
Not completed — Lost to Follow-up | 1 | 5 | 0 | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Includes all participants who started Stage 1
Groups:
- Resource Referral: Participants received a tailored list of information about community resources. The list will include information about local emergency food resources (e.g. local food pantries) and government programs to address food insecurity, such as the Supplemental Nutrition Assistance Program (SNAP).
- Community Health Worker (CHW) Intervention: Participants received assistance from a CHW. The CHW assisted participant with accessing community resources and worked with the patient's care team to assist with any barriers to care.
- Total: Total of all reporting groups
Arm/Group | Resource Referral | Community Health Worker (CHW) Intervention | Total
Number analyzed (Participants) | 28 | 32 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.3) | 58.1 (11.1) | 58.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 42
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 28 | 30 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 27 | 52
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Baseline Systolic Blood pressure [Mean (Standard Deviation); unit: mmHg] — Baseline blood pressure measured with ambulatory blood pressure monitor (mmHg)
  mmHg | 140.6 (10.1) | 151.8 (19.5) | 146.6 (16.7)
Baseline Diastolic Blood pressure [Mean (Standard Deviation); unit: mmHg] — Measured using ambulatory blood pressure monitor at baseline (mmHg)
  mmHg | 86.6 (9.9) | 88.4 (10.9) | 87.6 (10.4)

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure Readings
Description: assess blood pressure (using ambulatory blood pressure cuffs)
Time Frame: Baseline
Population: Participants in Stage 1 and Stage 2 arms
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Resource Referral + Community Health Worker (CHW) Intervention: This arm includes participants who did not respond to resource information in Stage 1. In Stage 1, participants received a tailored list of information about community resources. The list will include information about local emergency food resources (e.g. local food pantries) and government programs to address Food Insecurity (FI), such as the Supplemental Nutrition Assistance Program (SNAP).
  In Stage 2, nonresponders to resource information received assistance from a community health worker (CHW) for 3 months. The CHW helped participants with accessing community resources and worked directly with the patient's care team to assist with any barriers to care.
- Community Health Worker (CHW) + CHW Assistance: This arm includes participants who did not respond to CHW assistance in Stage 1. In Stage 1, participants received assistance from a CHW for 3 months. The CHW helped participants with access community resources and worked directly with the patients care team to assist with any barriers to care.
  In Stage 2, nonresponders to CHW assistance in Stage 1 received assistance from a CHW for an additional 3 months.
- Community Health Worker (CHW) Assistance + Medically Tailored Meals: This arm includes participants who did not respond to CHW assistance in Stage 1. In Stage 1, participants received assistance from a CHW for 3 months. The CHW helped participants with access community resources and worked directly with the patients care team to assist with any barriers to care.
  In Stage 2, nonresponders received 10 medically tailored meals delivered to their home weekly for 3 months.
Arm/Group | Resource Referral Only | Resource Referral + Community Health Worker (CHW) Intervention | Resource Referral + Medically Tailored Meals (MTM) | Community Health Worker (CHW) Only | Community Health Worker (CHW) + CHW Assistance | Community Health Worker (CHW) Assistance + Medically Tailored Meals
Number analyzed (Participants) | 13 | 7 | 8 | 18 | 6 | 8
mmHg | 144.3 (8.2) | 138.1 (9.1) | 136.8 (12.6) | 151.7 (18.2) | 150.8 (22.0) | 146.4 (16.1)

2. Primary Outcome: Feasibility of Recruitment Percentage
Description: Feasibility will be measured based on the proportion of patients screened who consented to be part of the study
Time Frame: Baseline
Population: 61 individuals screened met the inclusion and exclusion criteria. 60 individuals enrolled in the study and 1 declined
Measure: Number; unit: Proportion of participants
Groups:
- Proportion of Patients Who Consented to be Part of the Study: Feasibility will be measured based on the proportion of patients screened who consented to be part of the study
Arm/Group | Proportion of Patients Who Consented to be Part of the Study
Number analyzed (Participants) | 61
Proportion of participants | 0.98

3. Primary Outcome: Feasibility of Retention
Description: Feasibility will be measured at the proportion of participants who completed 3 and 6 month follow ups
Time Frame: Month 6
Population: Includes all participants who started Stage 1.
Measure: Number; unit: Proportion of participants
Groups:
- Resource Referral: Participants received a tailored list of information about community resources. The list will include information about local emergency food resources (e.g. local food pantries) and government programs to address Food Insecurity (FI), such as the Supplemental Nutrition Assistance Program (SNAP).
Arm/Group | Resource Referral | Community Health Worker (CHW) Intervention
Number analyzed (Participants) | 28 | 32
Proportion of participants | 0.5 | 0.625

4. Primary Outcome: Diastolic Blood Pressure Readings
Description: assess blood pressure (using ambulatory blood pressure cuffs)
Time Frame: Baseline
Population: Participants in Stage 1 and Stage 2 arms
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Resource Referral Only | Resource Referral + Community Health Worker (CHW) Intervention | Resource Referral + Medically Tailored Meals (MTM) | Community Health Worker (CHW) Only | Community Health Worker (CHW) + CHW Assistance | Community Health Worker (CHW) Assistance + Medically Tailored Meals
Number analyzed (Participants) | 13 | 7 | 8 | 18 | 6 | 8
mmHg | 87.4 (8.9) | 81.6 (8.1) | 89.8 (12.5) | 89.1 (11.5) | 88.3 (7.6) | 87.1 (12.7)

5. Primary Outcome: Systolic Blood Pressure Readings
Description: assess blood pressure (using ambulatory blood pressure cuffs)
Time Frame: Month 3
Population: 8 participants who started Stage 1 intervention did not complete 3 month follow-up (resource referral only arm) and 6 participants in the CHW only arm did not complete 3 month follow up
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Resource Referral Only | Resource Referral + Community Health Worker (CHW) Intervention | Resource Referral + Medically Tailored Meals (MTM) | Community Health Worker (CHW) Only | Community Health Worker (CHW) + CHW Assistance | Community Health Worker (CHW) Assistance + Medically Tailored Meals
Number analyzed (Participants) | 5 | 7 | 8 | 12 | 6 | 8
mmHg | 123.2 (12.1) | 165.8 (35.4) | 147.5 (12.5) | 124.7 (17.1) | 149.7 (20.1) | 171.6 (33.8)

6. Primary Outcome: Diastolic Blood Pressure Readings
Description: assess blood pressure (using ambulatory blood pressure cuffs)
Time Frame: Month 3
Population: 8 participants in the Resource referral only arm did not complete 3 month follow-up, 6 participants in the CHW only arm did not complete 3 month follow-up,
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Resource Referral Only | Resource Referral + Community Health Worker (CHW) Intervention | Resource Referral + Medically Tailored Meals (MTM) | Community Health Worker (CHW) Only | Community Health Worker (CHW) + CHW Assistance | Community Health Worker (CHW) Assistance + Medically Tailored Meals
Number analyzed (Participants) | 5 | 7 | 8 | 12 | 6 | 8
mmHg | 78.8 (10.4) | 103.6 (35.1) | 95.5 (6.6) | 79.0 (7.9) | 92.2 (22.3) | 103.8 (23.0)

7. Primary Outcome: Systolic Blood Pressure Readings
Description: assess blood pressure (using ambulatory blood pressure cuffs)
Time Frame: Month 6
Population: 1 participant in resource referral only arm did not complete 6 month follow-up, 5 participants in Resource referral + CHW arm did not complete 6 month follow-up, 3 participants in CHW only arm did not complete 6 month follow-up, 2 participants in CHW + CHW arm did not complete 6 month follow-up, and 1 participant in CHW + MTM arm did not complete follow-up
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Resource Referral Only | Resource Referral + Community Health Worker (CHW) Intervention | Resource Referral + Medically Tailored Meals (MTM) | Community Health Worker (CHW) Only | Community Health Worker (CHW) + CHW Assistance | Community Health Worker (CHW) Assistance + Medically Tailored Meals
Number analyzed (Participants) | 4 | 2 | 8 | 9 | 4 | 7
mmHg | 134.3 (23.2) | 158.2 (42.7) | 143.7 (22.9) | 138.3 (21.5) | 146.6 (13.5) | 158.7 (28.1)

8. Primary Outcome: Diastolic Blood Pressure Readings
Description: assess blood pressure (using ambulatory blood pressure cuffs)
Time Frame: Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Resource Referral Only | Resource Referral + Community Health Worker (CHW) Intervention | Resource Referral + Medically Tailored Meals (MTM) | Community Health Worker (CHW) Only | Community Health Worker (CHW) + CHW Assistance | Community Health Worker (CHW) Assistance + Medically Tailored Meals
Number analyzed (Participants) | 4 | 2 | 8 | 9 | 4 | 7
mmHg | 84.8 (16.0) | 116.3 (48.6) | 88 (12.4) | 86 (13.4) | 87.8 (12.3) | 98.0 (31.5)

ADVERSE EVENTS:
Time Frame: 6 Months
Groups:
- Resource Referral + CHW Intervention: This arm includes participants who did not respond to resource information in Stage 1. In Stage 1, participants received a tailored list of information about community resources. The list will include information about local emergency food resources (e.g. local food pantries) and government programs to address Food Insecurity (FI), such as the Supplemental Nutrition Assistance Program (SNAP).
  In Stage 2, nonresponders to resource information received assistance from a community health worker (CHW) for 3 months. The CHW helped participants with accessing community resources and worked directly with the patient's care team to assist with any barriers to care.
- Resource Referral + MTM: This arm included participants who did not respond to resource information in Stage 1. In Stage 1, participants received a tailored list of information about community resources. The list will include information about local emergency food resources (e.g. local food pantries) and government programs to address Food Insecurity (FI), such as the Supplemental Nutrition Assistance Program (SNAP).
  In Stage 2, nonresponders received 10 medically tailored meals delivered to their home weekly for 3 months.
- CHW + CHW Assistance: This arm includes participants who did not respond to CHW assistance in Stage 1. In Stage 1, participants received assistance from a CHW for 3 months. The CHW helped participants with access community resources and worked directly with the patients care team to assist with any barriers to care.
  In Stage 2, nonresponders to CHW assistance in Stage 1 received assistance from a CHW for an additional 3 months.
- CHW Assistance + MTM: This arm includes participants who did not respond to CHW assistance in Stage 1. In Stage 1, participants received assistance from a CHW for 3 months. The CHW helped participants with access community resources and worked directly with the patients care team to assist with any barriers to care.
  In Stage 2, nonresponders received 10 medically tailored meals delivered to their home weekly for 3 months.
Arm/Group | Resource Referral Only | Resource Referral + CHW Intervention | Resource Referral + MTM | Community Health Worker (CHW) Only | CHW + CHW Assistance | CHW Assistance + MTM
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/7 | 0/8 | 0/18 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/7 | 0/8 | 0/18 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/13 | 0/7 | 0/8 | 0/18 | 0/6 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT05800145/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT05800145/ICF_000.pdf